CLINICAL TRIAL: NCT06955442
Title: Analysis of Ethnic and Racial Disparities in Access to Acute Stroke Care in Italy: A Multicentric, Prospective Cohort Study
Brief Title: Racial Disparities in Acute Stroke
Acronym: ERDAS
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Frisullo Giovanni, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7467
Record Dates: First submitted 2025-04-16; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic Stroke; Health disparities; Equity in healthcare
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting to the ED for acute ischemic stroke: Patients will be divided into several subgroups based on their racial/ethnic belonging (Asian/Hispanic/Black/White/Others).

SUMMARY:
Ischemic stroke is one of the leading causes of mortality and disability worldwide. Although the prevalence of stroke is high globally, not all ethnic and racial groups are affected in the same way, leading to the classification of stroke as an inequitable disease.

First of all, ethnic and racial background influences the pathogenesis of stroke, as numerous risk factors-both modifiable and non-modifiable-are more prevalent in Black and Hispanic populations compared to Asian ones. As a direct consequence, the incidence of stroke is higher in Black and Hispanic individuals than in White individuals. Unfortunately, despite this, access to revascularization treatments is not always guaranteed for ethnic and racial minorities, although in recent years, this inequality in access to care appears to be decreasing.

Moreover, stroke prognosis also seems to differ based on race/ethnicity, with mortality being higher among Black individuals compared to White individuals, although this trend tends to decrease with advancing age. On the other hand, although cerebral hemorrhage is more prevalent in Black and Asian populations than in White populations, it tends to have a better prognosis in these minority groups.

It must be considered, however, that the vast majority of studies on this topic have been conducted in the United States, where the ethnic and racial composition of the population is very different from that of Italy and Europe. In these latter contexts, studies investigating the impact of race and/or ethnicity on the clinical characteristics, management, and prognosis of ischemic stroke are lacking. Furthermore, differences in healthcare system organization may play a significant role in limiting access to timely and appropriate medical care for acute stroke based on race and/or ethnicity.

Italy is a country where, similarly to other European nations, the last few decades have seen a significant increase in immigration rates, particularly from Eastern Europe. Today, foreigners account for approximately 9% of the total population. Nevertheless, in Italy, systemic racism toward ethnic and racial minorities remains a significant issue, as evidenced by large disparities in educational attainment, socioeconomic status, and housing conditions between Italian citizens and foreign residents.

Although the universal national healthcare system in Italy should ensure equal access to care and emergency treatment for all, regardless of ethnic and racial background, there are no studies investigating this topic. A recent scoping review highlighted how individual racism plays a primary role in generating health inequalities, whereas there is very limited evidence focused on the analysis of structural and institutional racism in the Italian and European context.

As a consequence, this study aims to prospectively investigate the presence and the extent of racial and ethnic disparities in access to stroke care and treatment across several Italian comprehensive stroke centers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old);
* Admission to the Emergency Department of the participating center with a diagnosis of ischemic stroke, as defined by the International Classification of Diseases, 9th Revision (ICD-9) codes;
* Signed informed consent provided by the patient or, in cases of impaired decision-making capacity, by their legal guardian/representative.

Exclusion Criteria:

* Discharge diagnosis other than ischemic stroke;
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED of a hospital for a suspected stroke diagnosis. Patients will be then divided into different subgroups according to their racial/ethnic belonging (White, Asian, Hispanic, Black, Others).
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Racial/ethnic disparities in the access to revascularization treatments | Baseline
  Comparison of the likelihood of undergoing revascularization treatments among patients from different racial and/or ethnic groups.

SECONDARY OUTCOMES:
Racial/ethnic disparities in onset to door times | Baseline
  Comparison of Onset-to-Door Time among patients from different racial and/or ethnic groups.
Racial/ethnic disparities in door to needle times | From the time of ED admission at baseline to start of intravenous thrombolysis
  Comparison of differences in Door-to-Needle Time (DTN) between patients from different racial and/or ethnic groups.
Racial/ethnic disparities in door to groin times | From the time of ED admission at baseline to femoral puncture for mechanical thrombectomy
  Comparison of differences in Door-to-Groin Time (DTG) between patients from different racial and/or ethnic groups.
Racial/ethnic differences in mode of emergency department arrival | Baseline
  Comparison of ED arrival modes (walk-in vs emergency medical services) among patients from different racial and/or ethnic groups.
Racial/ethnic differences in the prevalence of cardiovascular risk factors | Baseline
  Comparison of the prevalence of cerebrovascular risk factors among patients from different racial and/or ethnic groups.
Racial/ethnic differences in onset symptoms of stroke | Baseline
  Comparison of stroke clinical presentation patterns among patients from different racial and/or ethnic groups.
Racial/ethnic differences in stroke pathogenesis | From enrollment to hospital discharge, up to 90-days from baseline
  Comparison of stroke etiologies, classified according to the Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria, among patients from different racial and/or ethnic groups.
Racial/ethnic differences stroke outcome at discharge | From enrollment to hospital discharge, up to 90-days from baseline
  Comparison of discharge modified Rankin Scale (mRS) scores among patients from different racial and/or ethnic groups.
Racial/ethnic differences in 3-month stroke outcome | From enrollment to the 3-month follow-up visit
  Comparison of 3-month modified Rankin Scale (mRS) scores after acute ischemic stroke among patients from different racial and/or ethnic groups.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Frisullo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (15):
- Italy (15):
  - Ospedale Maggiore, IRCCS Istituto delle Scienze Neurologiche di Bologna - UO Neurologia OM e Rete Stroke Metropolitana (SC), Bologna
  - UOS Neurologia-AOU, IRCCS Istituto delle scienze Neurologiche, Bologna
  - UOC Neurologia, ASST Crema, Crema
  - UOC Neurologia - Ospedale Spaziani, Frosinone
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale Vito Fazzi, Lecce
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Naples
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - IRCCS Fondazione Istituto Neurologico C. Mondino, Pavia
  - IRCCS Istituto Neurologico Mediterraneo Neuromed, Pozzilli
  - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I, Rome
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
  - Humanitas Research Hospital IRCCS, Rozzano
  - UOC Neurologia Belcolle - Ospedale Belcolle, Viterbo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frisullo G, Scala I, Di Giovanni J, Rizzo PA, Bellavia S, Broccolini A, Monforte M, Franceschi F, Gasbarrini A, Carbone L, Calabresi P, Covino M. Racial and ethnic differences in access to care and treatment in patients with suspected acute stroke: A retrospective, observational, cohort study. J Neurol Sci. 2024 Nov 15;466:123225. doi: 10.1016/j.jns.2024.123225. Epub 2024 Sep 10. PMID 39270410

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT06955442/Prot_SAP_000.pdf